CLINICAL TRIAL: NCT01394393
Title: Ambientes Virtuales Como Auxiliares en el Tratamiento de la Obesidad
Brief Title: Virtual Environments For Supporting Obesity Treatment
Acronym: AVATOB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Istituto Auxologico Italiano (Other); Medica Sur Clinic & Foundation (Other)
Responsible Party: Principal Investigator, DRA. GEORGINA CARDENAS LOPEZ, Full time professor, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SALUD-2010-1-140220; SALUD-2010-1-140220.PHASE1 (Other: UNIVERSIDAD NACIONAL AUTONOMA DE MEXICO)
Record Dates: First submitted 2011-06-27; First posted 2011-07-14 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Obesity; Morbid Obesity
Keywords: obesity treatment; evidence based intervention; cognitive behavioral treatment; virtual reality environments
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Adiposity; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ECT (Experimental): Experiential-Cognitive Therapy for Obesity
  Interventions: Behavioral: Experiential-Cognitive Therapy for Obesity
- BCT (Active Comparator): Cognitive behavioral treatment program
  Interventions: Behavioral: Behavioral cognitive Treatment
- NT (Sham Comparator): Nutritional groups In this condition (NT) the participants enter only 5 weekly nutritional groups held by dietitians.
  Interventions: Dietary Supplement: Nutritional groups (NT)

INTERVENTIONS:
Behavioral: Experiential-Cognitive Therapy for Obesity — Is a relatively short-term, integrated, patient oriented approach that focuses on individual discovery (Riva, Bacchetta, Baruffi, Rinaldi, & Molinari, 1998, 1999; Riva et al., 2000). It shares with the cognitive-behavioral approach proposed by Cooper and colleagues the use of a combination of cognitive and behavioral procedures to help the patient identify and change the maintaining mechanisms (Cooper et al., 2003). However, it considers morbid obesity as a peculiar form of addiction. So, as in the cognitive-behavioral treatment of addictions (Carroll et al., 1994) the two main goals are the functional analysis of the maintaining mechanisms and the required skill training (relapse prevention).
  Other Names: Virtual Reality Enhanced Therapy for Obesity
  Arms: ECT
Behavioral: Behavioral cognitive Treatment — Therapists will follow a detailed manual that outlined the content of each session. This manual was based on the cognitive-behavioral treatment approach described by Cooper and colleagues (Cooper & Fairburn, 2002; Cooper et al., 2003). It was developed during a year of intensive pilot work and adapted to the in-patient setting. Patients will be taught to self-monitor their food intake and eating patterns and thoughts, as well as the circumstances and environment surrounding eating (e.g. whether eating alone or with others, speed of eating, and place of eating). Patients will also be taught to identify problems in eating, mood, and thinking patterns and to gradually develop alternative patterns.
  Other Names: Behavioral cognitive therapy; Obesity cognitive behavioral approach
  Arms: BCT
Dietary Supplement: Nutritional groups (NT) — 5 weekly nutritional treatment based on the LEARN manual (Brownell, 1985), whose goal will be to provide practical guidelines for the self-monitoring of eating and lessons on nutrition (e.g stressing gradual weight loss with the caloric restriction achieved largely by reductions in fat intake), plus a low-calorie diet (1,200 kcal/day) and physical training (30 min of walking two times a week as a minimum).
  Other Names: Nutritional treatment
  Arms: NT

SUMMARY:
Participants 60 Patients seeking treatment at the Obesity Unit of the Medica Sur Hospital in México City, Mexico. Informed consent to participate will be aleatory assigned to a three different conditions.

Procedures In the initial interview, prospective participants will be provided with detailed information about the study and the treatments. All patients included in the study will be randomly assigned to the one (N=20) of the three treatment conditions described below, all conducted on an inpatient basis. The duration for all treatments will be 6 weeks and will be administered by two chartered clinical psychologists and one chartered psychotherapist under the supervision of a senior chartered psychotherapist. The three therapists will be balanced among the three conditions.

1. Nutritional groups In this condition (NT) the participants (N=20) subjects enter only 5 weekly nutritional groups held by dieticians based on the LEARN manual (Brownell, 1985), whose goal will be to provide practical guidelines for the self-monitoring of eating and lessons on nutrition (e.g stressing gradual weight loss with the caloric restriction achieved largely by reductions in fat intake), plus a low-calorie diet (1,200 kcal/day) and physical training (30 min of walking two times a week as a minimum).
2. Cognitive-Behavioral therapy CBT group (N=20) will be based on the same treatment proposed in the first condition plus 15 additional sessions over 6 weeks.

   Therapists will follow a detailed manual that outlined the content of each session. This manual was based on the cognitive-behavioral treatment approach described by Cooper and colleagues (Cooper & Fairburn, 2002; Cooper et al., 2003). It was developed during a year of intensive pilot work and adapted to the in-patient setting. Patients will be taught to self-monitor their food intake and eating patterns and thoughts, as well as the circumstances and environment surrounding eating (e.g. whether eating alone or with others, speed of eating, and place of eating). Patients will also be taught to identify problems in eating, mood, and thinking patterns and to gradually develop alternative patterns.

   In particular, after the first week the patients will enter 5 weekly group sessions aimed at addressing weight and primary goals, and 10 biweekly individual sessions aimed at establishing and maintaining weight loss, addressing barriers to weight loss, increasing activity, addressing body image concerns and supporting weight maintenance.
3. Experiential Cognitive therapy Experiential CT group (N=4) involved the same treatment proposed in the first condition plus 15 additional sessions over 4/6 weeks.

In the sessions we will use the "20/20/20 rule". During the first 20 minutes, the therapist focus on getting a clear understanding of the patient's current concerns, level of general functioning, and the experiences related to food. This part of the session tends to be characterized by patients doing most of the talking, although therapist guides with questions and reflection to get a sense of the patient's current status. The second 20 minutes is devoted to the virtual reality experience. During this part of the session the patient enters the virtual environment and faces a specific critical situation (Kitchen, Supermarket, Pub, Restaurant, Gymnasium, etc.). Here the patient is helped in developing specific strategies for avoiding and/or coping with it. In the final 20 minutes the therapist explores the patient's understanding of what happened in VR and the specific reactions - emotional and behavioral - to the different situations experienced. If needed, some new strategies for coping with the VR situations are presented and discussed. To support the empowerment process, the therapists follow the Socratic style: they use a series of questions, related to the contents of the virtual environment, to help clients synthesize information and reach conclusions on their own.

In accordance with informed consent, assessments will be obtained before treatment, at posttreatment, 3 and 6 months after the treatment conclusion.

DETAILED DESCRIPTION:
In the initial interview, prospective participants will be provided with detailed information about the study and the treatments. All patients included in the study will be randomly assigned to the waiting-list group and to the one of the three treatment conditions described below, all conducted on an inpatient basis. The duration for all treatments will be 6 weeks and will bw administered by two chartered clinical psychologists and one chartered psychotherapist under the supervision of a senior chartered psychotherapist. The three therapists will bw balanced among the three conditions. In accordance with informed consent, assessments will be obtained before treatment, at posttreatment, 3 and 6 months follow up after the end of treatment.

1. Nutritional groups In this condition (NT) the subjects enter only 5 weekly nutritional groups held by dieticians based on the LEARN manual (Brownell, 1985), whose goal will be to provide practical guidelines for the self-monitoring of eating and lessons on nutrition (e.g stressing gradual weight loss with the caloric restriction achieved largely by reductions in fat intake), plus a low-calorie diet (1,200 kcal/day) and physical training (30 min of walking two times a week as a minimum).

2 Cognitive-Behavioral therapy CBT will be based on the same treatment proposed in the first condition plus 15 additional sessions over 6 weeks. Therapists will follow a detailed manual that outlined the content of each session. This manual was based on the cognitive-behavioral treatment approach described by Cooper and colleagues (Cooper & Fairburn, 2002; Cooper et al., 2003). It was developed during a year of intensive pilot work and adapted to the in-patient setting. Patients will be taught to self-monitor their food intake and eating patterns and thoughts, as well as the circumstances and environment surrounding eating (e.g. whether eating alone or with others, speed of eating, and place of eating). Patients will also be taught to identify problems in eating, mood, and thinking patterns and to gradually develop alternative patterns. In particular, after the first week the patients will enter 5 weekly group sessions aimed at addressing weight and primary goals, and 10 biweekly individual sessions aimed at establishing and maintaining weight loss, addressing barriers to weight loss, increasing activity, addressing body image concerns and supporting weight maintenance.

3. Experiential Cognitive therapy In particular, after the first week the patients entered 5 weekly group sessions aimed at improving motivation to change and assertiveness, and 10 biweekly virtual reality sessions. For the VR sessions, the NeuroVR 1.5 software will be used. NeuroVR is an enhanced version of the original Virtual Reality for Body Image Modification (VEBIM) immersive virtual environment, previously used in different preliminary studies on non-clinical subjects (Riva, 1997a, 1998b). Is composed of 14 virtual environments, used by the therapist within a 60-minute session with the patient. The environments present critical situations related to the maintaining/relapse mechanisms (Home, Supermarket, Pub, Restaurant, Swimming Pool, Beach, Gymnasium) and two body image comparison areas.

Using the NeuroVR Editor, the psychological stimuli/stressors appropriate for any given scenario can be chosen from a rich database of 2D and 3D objects, and easily placed into the pre-designed virtual scenario by using an icon-based interface (no programming skills are required). In addition to static objects, the NeuroVR Editor allows both to add audio object and to overlay on the 3D scene video composited with a transparent alpha channel.The editing of the scene is performed in real time, and effects of changes can be checked from different views (frontal, lateral and top).

The edited scene is then visualized and experienced using the NeuroVR Player. Through the VR experience, the patients practice both eating/emotional/relational management and general decision-making and problem-solving skills. By directly practicing these skills within the VR environment, the patient is helped in developing specific strategies for avoiding and/or coping with these.

9 sessions are used to assess and modify:

* the expectations and emotions related to food and weight: This is done both by integrating different cognitive-behavioral methods: Countering, Alternative Interpretation, Label Shifting, Deactivating the Illness Belief
* the strategies used to cope with difficult interpersonal and potential maintenance situations: This is done both by using the Temptation Exposure with Response Prevention (Riva, 1998c; D. G. Schlundt & Johnson, 1990) - and by working on these three empowering dimensions (Menon, 1999): perceived control, perceived competence and goal internalization.
* the body experience of the subject. To do this the virtual environment integrates the therapeutic methods used by Butter & Cash (1987) and Wooley & Wooley (1985). In particular in VREDIM we used the virtual environment in the same way as guided imagery (Leuner, 1969) is used in the cognitive and visual/motorial approach.

Structure of the sessions

Each session of Virtual Reality is divided into four phases:

The psychologist's office is the first virtual experience. It represents the start and the end of each session, and it has the important function to outline boundaries of the session in virtual reality. It is a neutral and reassuring place which allows continuity in the phases of the individual session: face to face, virtual reality and face to face.

In the psychologist's office there are the following objects: a writing-desk with two comfortable chairs, a bookshelf and complements of furnishings that make the environment more comfortable and hospitable (pictures, carpets, lamps, green plants, etc.). The safe place is the virtual experience for the relaxation that is used at the end of each session and, if needed, during the session of virtual reality. It is an empty park in which the patient can relax and recover from any emotional experience.

Between the psychologist's office and the safe place the patient experiences one or more specific virtual experience.

In accordance with informed consent, assessments will be obtained before treatment, at posttreatment, 3 and 6 months after the treatment conclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients seeking treatment at the Obesity Unit of the Hospital Medica Sur, Mexico City, Mexico
2. a Body Mass Index higher than 40;
3. written and informed consent to participate.

Exclusion Criteria:

1. other concurrent severe psychiatric disturbances (psychosis, depression with suicidal risk, alcohol or drug abuse);
2. concurrent medical condition not related to the disorder;
3. one or more failures in following an obesity treatment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety Inventory: State-Trait IDARE | Change from Baseline in Anxiety Inventory: State-Trait IDARE at 6 weeks, Change from Baseline in Anxiety Inventory: State-Trait IDARE at 6 months
  The scale A-Trait Anxiety Inventory consists of twenty statements in which subjects are asked to describe how they feel generally. A-State scale also consists of 20 statements, but the instructions required that subjects indicate how they feel at any given time. Measures two dimensions of anxiety: state (referring to how the subject feels at that moment) and trait (how you feel usually). Instrument validated in Mexico (Spielberger & Diaz Guerrero, 1975)
Body Image Questionnaire (BSQ) | Change frome Baseline in Body Image Questionnaire (BSQ) at 6 weeks, Change frome Baseline in Body Image Questionnaire (BSQ) at 6 months
  Designed by Cooper, Taylor, Cooper and Fairburn (1987), adapted to Spanish population by Raich et al. (1996) and to Mexican women by Galán (2004). Consists of 34 questions scored on a Likert scale of 1 to 6. Lets get an overall score (sum of raw scores of the items) and can be derived 4 subscales: body dissatisfaction, fear of gaining weight, low esteem by the appearance and want to lose weight.
Weight | Changes in weight from de first week will be assessed up to 6 weeks, changes in weight at 6 months
  Weight loss after the treatment and after the follow-up phase

SECONDARY OUTCOMES:
BULIT Bulimia Test | Change from Baseline in BULIT Bulimia Test at 6 weeks, Change from Baseline in BULIT Bulimia Test at 6 months
  Self-administered questionnaire of 36 items designed to assess bulimic symptomatology (Smith & Thelen, 1984). The questions are related to body weight, binge mood and purgative behavior. Adapted to Mexican population (Alvarez & Vazquez-Manzilla, 2000).
Three Food Factors Questionnaire (TFEQ) | Change from Baseline in Three Food Factors Questionnaire (TFEQ) at 6 weeks, Change from Baseline in Three Food Factors Questionnaire (TFEQ) at 6 months
  Questionnaire comprising 51 items that measure three factors: cognitive dietary restraint, ie the perception that food intake is limited constants in an effort to control the body weight, disinhibition and hunger. (Stunkard & Messick, 1985).
Opinion on exposure therapy | Opinion on exposure therapy at 6 weeks
  Questionnaire developed for this study, which will reflect the level of satisfaction with treatment, which will assess how useful it has been each of the components of the treatment program (educational component, relaxation training, exposure component of each virtual scenarios (for conditions with virtual reality exposure).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Riva, PhD, Study Chair — Catholic University of Milan; Gonzalo Torres-Villalobos, MD, Study Director — Medica Sur Foundation; Andrea Gaggioli, PhD, Study Director — Istituto Auxologico Italiano
Locations (1):
- Hospital Medica Sur, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Riva G, Bacchetta M, Cesa G, Conti S, Castelnuovo G, Mantovani F, Molinari E. Is severe obesity a form of addiction? Rationale, clinical approach, and controlled clinical trial. Cyberpsychol Behav. 2006 Aug;9(4):457-79. doi: 10.1089/cpb.2006.9.457. PMID 16901250
- [Background] Riva G, Bacchetta M, Baruffi M, Molinari E. Virtual reality-based multidimensional therapy for the treatment of body image disturbances in obesity: a controlled study. Cyberpsychol Behav. 2001 Aug;4(4):511-26. doi: 10.1089/109493101750527079. PMID 11708731
- [Background] Riva G. The key to unlocking the virtual body: virtual reality in the treatment of obesity and eating disorders. J Diabetes Sci Technol. 2011 Mar 1;5(2):283-92. doi: 10.1177/193229681100500213. PMID 21527095
- See also: A previous Italian controlled trial based on the same protocol (it also included eating disorders, not covered by the actual trial) — http://www.controlled-trials.com/ISRCTN59019572